CLINICAL TRIAL: NCT00462709
Title: LEVP2006-4 CHANGE 3 Trial (C1-Inhibitor in Hereditary Angioedema Nanofiltration Generation Evaluating Efficacy): Open-Label Use of C1INH-nf (Human) for the Prophylactic Treatment to Prevent HAE Attacks and as Treatment in Acute HAE Attacks
Brief Title: Open-Label C1 Esterase Inhibitor (C1INH-nf) for the Prevention of Acute Hereditary Angioedema (HAE) Attacks
Acronym: CHANGE 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LEVP2006-4
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2010-05-03 (Estimated); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary angioedema; C1 esterase inhibitor (human)
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein

ARMS (1):
- Open-label C1INH-nf (Experimental): 1,000 Units (U) of C1INH-nf administered intravenously (IV) every 3 to 7 days.
  Interventions: Biological: C1 esterase inhibitor [human] (C1INH-nf)

INTERVENTIONS:
Biological: C1 esterase inhibitor [human] (C1INH-nf)

SUMMARY:
The study objective was to evaluate the safety and efficacy of prophylactic use of C1INH-nf for the prevention of acute HAE attacks.

ELIGIBILITY:
Inclusion Criteria:

- History of at least 1 HAE attack per month or any history of laryngeal edema

In addition, this study was open to all subjects who:

* Completed participation in LEVP2005-1/B (NCT01005888) any time after the final prophylactic therapy in Part B
* Were enrolled but not randomized in LEVP2005-1/A (NCT00289211) after Part A was closed
* Were enrolled and randomized in LEVP2005-1/A after LEVP2005-1/B was closed to enrollment, any time after the 3-day telephone follow-up
* Were excluded from LEVP2005-1 for any of the following reasons:

  * Pregnancy or lactation
  * Age less than 6 years
  * Narcotic addiction
  * Presence of anti-C1 inhibitor (C1INH) autoantibodies
* Were not enrolled in LEVP2005-1 after enrollment in LEVP2005-1 was closed, under the following circumstances:

  * Had a diagnosis of HAE: evidence of a low C4 level plus either a low C1INH antigenic level or a low C1INH functional level, or
  * Had a known HAE-causing C1INH mutation, or
  * Had a diagnosis of HAE based on a strong family history of HAE as determined by the principal investigator

Exclusion Criteria:

* History of allergic reaction to C1INH or other blood products
* Participated in any other investigational drug study within the past 30 days other than those sponsored by Lev Pharmaceuticals
* Received blood or a blood product in the past 60 days other than C1INH-nf

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2006-06-27 (Actual); Primary Completion 2009-03-31 (Actual); Study Completion 2009-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (48):
- United States (48):
  - Clinical Research Consultants, Inc, Hoover, Alabama
  - Allergy and Immunology Associates, Scottsdale, Arizona
  - Allergy and Asthma Clinic of Northwest Arkansas, Bentonville, Arkansas
  - UCLA-David Geffen School of Medicine, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Allergy and Asthma Associates of Santa Clara, San Jose, California
  - Allergy and Asthma Clinical Research, Inc, Walnut Creek, California
  - Allergy and Asthma Center, Fort Lauderdale, Florida
  - Allergy and Asthma Center of East Orlando, Orlando, Florida
  - Cleveland Clinic, Weston, Florida
  - Family Allergy and Asthma Center, Atlanta, Georgia
  - Atlanta Allergy and Asthma Clinic, Suwanee, Georgia
  - University Consultants in Allergy & Immunology, Chicago, Illinois
  - Welborn Clinic, Evansville, Indiana
  - Private Practice, Liberal, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Family Asthma and Allergy Research Center, Louisville, Kentucky
  - Asthma Allergy and Sinus Center, Waldorf, Maryland
  - Institute for Asthma and Allergy, Wheaton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Grand Traverse Allergy, Traverse City, Michigan
  - MeritCare Clinical Research, Bemidji, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis University School of Medicine, St Louis, Missouri
  - Nevada Access to Research and Education Society, Las Vegas, Nevada
  - UMDNJ Asthma and Allergy Research Center, Newark, New Jersey
  - Private Practice, Hastings-on-Hudson, New York
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai School of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Allergy Partners of East Carolina, Greenville, North Carolina
  - Legacy Pharma Research, Bismarck, North Dakota
  - MeritCare Clinical Research, Fargo, North Dakota
  - Nationwide Childrens Hospital Clinical Research, Columbus, Ohio
  - Allergy Clinic of Tulsa, Tulsa, Oklahoma
  - Oregon Medical Group, Eugene, Oregon
  - Allergy Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - Penn State University, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - Pediatric Pulmonary/Allergy and Immunology, Houston, Texas
  - Allergy and Asthma Research Center, San Antonio, Texas
  - Tyler County Hospital, Woodville, Texas
  - Virginia Adult and Pediatric Allergy and Asthma, Richmond, Virginia
  - Marycliff Allergy Specialists, Spokane, Washington
  - Puget Sound Allergy, Asthma and Immunology, Tacoma, Washington
  - St. Joseph's Hospital/Cornerstone Healthcare, Parkersburg, West Virginia

REFERENCES:
- [Derived] Beard N, Frese M, Smertina E, Mere P, Katelaris C, Mills K. Interventions for the long-term prevention of hereditary angioedema attacks. Cochrane Database Syst Rev. 2022 Nov 3;11(11):CD013403. doi: 10.1002/14651858.CD013403.pub2. PMID 36326435
- [Derived] Baker JW, Craig TJ, Riedl MA, Banerji A, Fitts D, Kalfus IN, Uknis ME. Nanofiltered C1 esterase inhibitor (human) for hereditary angioedema attacks in pregnant women. Allergy Asthma Proc. 2013 Mar-Apr;34(2):162-9. doi: 10.2500/aap.2013.34.3645. PMID 23484892
- [Derived] Lumry W, Manning ME, Hurewitz DS, Davis-Lorton M, Fitts D, Kalfus IN, Uknis ME. Nanofiltered C1-esterase inhibitor for the acute management and prevention of hereditary angioedema attacks due to C1-inhibitor deficiency in children. J Pediatr. 2013 May;162(5):1017-22.e1-2. doi: 10.1016/j.jpeds.2012.11.030. Epub 2013 Jan 11. PMID 23312695
- [Derived] Zuraw BL, Busse PJ, White M, Jacobs J, Lumry W, Baker J, Craig T, Grant JA, Hurewitz D, Bielory L, Cartwright WE, Koleilat M, Ryan W, Schaefer O, Manning M, Patel P, Bernstein JA, Friedman RA, Wilkinson R, Tanner D, Kohler G, Gunther G, Levy R, McClellan J, Redhead J, Guss D, Heyman E, Blumenstein BA, Kalfus I, Frank MM. Nanofiltered C1 inhibitor concentrate for treatment of hereditary angioedema. N Engl J Med. 2010 Aug 5;363(6):513-22. doi: 10.1056/NEJMoa0805538. PMID 20818886

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label C1INH-nf: 1,000 Units (U) of C1 esterase inhibitor (C1INH-nf) administered intravenously (IV) every 3 to 7 days.
Period: Overall Study
Arm/Group | Open-label C1INH-nf
Started | 146
Completed | 79
Not Completed | 67
Not completed — Transitioned to commercial C1INH-nf | 40
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 8
Not completed — Transferred to LEVP2006-1 (NCT00438815) | 3
Not completed — Death | 2
Not completed — Logistical reasons | 2
Not completed — Physician Decision | 1
Not completed — Withdrew to start treatment with Cetor | 1

BASELINE CHARACTERISTICS:
Groups:
- Open-label C1INH-nf: 1,000 U of C1INH-nf administered IV every 3 to 7 days.
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (16.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Frequency of All HAE Attacks
Description: A hereditary angioedema (HAE) attack was defined as a discrete episode during which the subject progressed from no angioedema to symptoms of angioedema.
Time Frame: Duration of the study
Population: Intent-to-treat Efficacy (ITT-E) Population (N=146; the number of subjects who received at least one prophylactic dose of C1INH-nf for the prevention of HAE attacks). HAE attack frequency was reported by 137 subjects at screening (i.e., data were missing for 9 subjects).
Measure: Median (Full Range); unit: attacks per month
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 146
attacks per month
  At Screening (N=137) | 3.00 [0.08 to 28.00]
  During Prophylactic Therapy with C1INH-nf (N=146) | 0.21 [0.00 to 4.56]

2. Other Pre Specified Outcome: Antigenic C1 Inhibitor (C1INH) Serum Levels
Description: Change from pre-infusion to 1 hour post-infusion in antigenic C1INH serum levels.
Time Frame: Pre-infusion to 1 hour post-infusion
Population: ITT-E subjects with data at both sampling time points (N=137).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 137
mg/dL
  Pre-infusion | 17.1 (19.67)
  Increase at 1 hour post-infusion | 8.6 (11.89)

3. Other Pre Specified Outcome: Functional C1INH Serum Levels
Description: Change from pre-infusion to 1 hour post-infusion in functional C1INH serum levels. Functional C1INH serum levels are expressed as a percent of total detectable C1INH (i.e., functional C1INH/total detectable C1INH).
Time Frame: Pre-infusion to 1 hour post-infusion
Population: ITT-E subjects with data at both sampling time points (N=132).
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 132
percent
  Pre-infusion | 42.0 (25.85)
  Percent increase at 1 hour post-infusion | 30.4 (18.05)

4. Other Pre Specified Outcome: Complement C4 Serum Levels
Description: Change from pre-infusion to 1 hour post-infusion in complement C4 serum levels.
Time Frame: Pre-infusion to 1 hour post-infusion
Population: ITT-E subjects with data at both sampling time points (N=134).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open-label C1INH-nf
Number analyzed (Participants) | 134
mg/dL
  Pre-infusion | 10.1 (8.17)
  Change at 1 hour post-infusion | -0.1 (3.61)

ADVERSE EVENTS:
Description: Presented are treatment-emergent adverse reactions considered to be related to C1INH-nf. There were no serious adverse reactions considered related to C1INH-nf.
Arm/Group | Open-label C1INH-nf
Serious Adverse Events (participants affected / at risk) | 0/146
Other Adverse Events (participants affected / at risk) | 9/146
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label C1INH-nf (N=146)
Nausea (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Phlebitis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Clinical Study Agreement. Most restrictive provision - PI will not publish results until after first of: multicenter publication is published or 24 months from study end. Thereafter, PI may publish his results. PI must provide copy of proposed publication to sponsor for pre-review. If sponsor requests, PI must delete sponsor confidential information before publication and/or delay publication for 90 days so sponsor can file for patents or take other action to protect its patent rights.